CLINICAL TRIAL: NCT05934240
Title: The Immediate Effect of Manual Therapy Application on Respiratory Functions in Healthy
Brief Title: The Immediate Effect of Manual Therapy Application on Respiratory Functions in Healthy Young Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Eylem KÜÇÜK, Lecturer, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: HacettepeUEKC
Record Dates: First submitted 2023-06-21; First posted 2023-07-06 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Health Young Individuals
Keywords: Manual therapy; Respiratory function test; Physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Active Comparator): Diaphragmatic mobilization, toracic mobilization and manipulation
  Interventions: Other: Manual therapy group
- Control group (Placebo Comparator): Placebo mobilization and manipulation
  Interventions: Other: Sham-manual therapy

INTERVENTIONS:
Other: Manual therapy group — Manual therapy will be applied to the diaphragm and thoracic region.
  Arms: Experimental group
Other: Sham-manual therapy — Sham-manual therapy will be applied to the diaphragm and thoracic region.
  Arms: Control group

SUMMARY:
Manual therapy techniques targeting the thoracic region are commonly used in clinical practice. It has been suggested that manual therapy interventions directed at the spine can increase mobility of the spine and chest wall, which may have a positive impact on lung functions. The potential positive effects of thoracic manipulation on respiratory system diseases such as chronic obstructive pulmonary disease (COPD) and asthma have been investigated and continue to be studied. Specifically, the results of studies investigating the physiological outcomes of this therapeutic approach in healthy adults are conflicting. The aim of this study is to investigate the short-term effects of thoracic manipulation and mobilization, as well as diaphragm mobilization, through a single session of manual therapy interventions on respiratory functions.

DETAILED DESCRIPTION:
In this planned study, designed as a randomized controlled intervention trial, two groups will be formed: an experimental group and a control group. After completing these procedures, the intervention group will receive the method of "thoracic mobilization and manipulation with diaphragm mobilization," while the control group will receive a placebo thoracic mobilization method. All techniques will be applied by a physiotherapist.

Within 5 minutes after the completion of the intervention, a respiratory function test will be repeated, resulting in a total of two respiratory function tests: one before the intervention and one after the intervention. The changes in respiratory function criteria before and after the intervention will be compared in both groups

ELIGIBILITY:
Inclusion Criteria:

* be between the ages of 18-25,
* to be a studen

Exclusion Criteria:

* those who have any health problems
* those with orthopedic disorders
* those with systemic and cardiopulmonary diseases that would interfere with the evaluation

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Pulmonary Functions Test- FEV1 (Forced expiratory volume in the first second) | Change from before and 5 minutes after application
  The forced expiratory volume in 1 second (FEV1) is the volume of air (in liters) exhaled in the first second during forced exhalation after maximal inspiration.
Pulmonary Functions Test-FVC (Forced vital capacity) | Change from before and 5 minutes after application
  Forced vital capacity, the maximum amount of air you can forcibly exhale from your lungs after fully inhaling.
Pulmonary Functions Test- FEV1/FVC | Change from before and 5 minutes after application
  The FEV1/FVC ratio is the ratio of the forced expiratory volume in the first one second to the forced vital capacity of the lungs.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Kucuk E, Tozcu D, Topaktas B, Coskun G. Immediate effects of manual therapy on respiratory functions in healthy young individuals: a randomized controlled trial. Sci Rep. 2024 Jul 29;14(1):17419. doi: 10.1038/s41598-024-68654-7. PMID 39075156